CLINICAL TRIAL: NCT04749823
Title: The NEXERCISE-trial: When Pain Neuroscience and Clinical Exercise Physiology Meet: Reshaping Exercise Programs for Patients With Non-specific Neck Pain
Brief Title: The NEXERCISE-trial: Reshaping Exercise Programs for Patients With Non-specific Neck Pain
Acronym: NEXERCISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-5419
Record Dates: First submitted 2020-10-26; First posted 2021-02-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Neck Pain; Chronic Pain
Keywords: local neck exercises; general aerobic exercises; pain intensity; cost effectiveness
MeSH Terms: conditions — Neck Pain; Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blended treatment program (Experimental): The blended treatment program will consist of a combination of specific active exercises of the neck and general aerobic exercises. This contains a program of 12 weeks, including 9 supervised online sessions supplemented with 1 to 3 individual home exercises sessions without supervision per week, with a total of 3 sessions/week.
  Interventions: Other: Blended treatment program
- Specific strength exercise program (Active Comparator): This group will receive an exercise program with specific strength exercises of the neck muscles. Within a 12-week period, patients will receive 9 online treatment sessions under supervision and 1 to 3 additional home exercise sessions without supervision, with a total of 3 sessions/week..
  Interventions: Other: Specific strength exercise program
- General aerobic exercise program (Active Comparator): This control group will perform general aerobic exercises. Within a 12-week period, patients will be instructed to perform a general aerobic exercise session 3 times a week.
  Interventions: Other: General aerobic exercise program

INTERVENTIONS:
Other: Blended treatment program — A combined treatment program with specific active neck exercises and general aerobic training in counteractive amount will be executed during 12 weeks. Nine supervised sessions will be supplemented with 1 to 3 weekly unsupervised home exercise sessions.
  Arms: Blended treatment program
Other: Specific strength exercise program — This program includes an individual, patient-tailored exercise program with the aim of retraining the neck musculature. A detailed exercise programme will be constructed in which all exercises are listed with the amount of repetitions and series of each exercise. Strength exercises will be performed by means of dumbbells with different weights and elastic bands with different degrees of resistance. The amount of weight or resistance, and the amount of series and repetitions will be evaluated during the first session. This exercise programme will be re-evaluated repeatedly during the course of the program. Specific strength neck exercises will be performed for 30 minutes. Nine supervised sessions will be supplemented with 1 to 3 weekly unsupervised home exercise sessions.
  Arms: Specific strength exercise program
Other: General aerobic exercise program — This control group will receive a general aerobic exercise program. Within a 12-week period, patients will be instructed to perform a general aerobic exercise session 3 times a week.
  Arms: General aerobic exercise program

SUMMARY:
The Nexercise-trial is a blended treatment program for patients with chronic non-specific neck pain. We will investigate whether a blended treatment approach, combining specific neck exercises and general aerobic exercises, has better outcome (on medical impact for the patient and socio-economic impact) than a specific neck exercise program alone or a general aerobic exercise program alone.

DETAILED DESCRIPTION:
Chronic non-specific neck pain is a common musculoskeletal complaint in which several biopsychosocial factors can be involved. This condition is associated with a high socio-economic burden. The standard of care treatment for chronic neck pain in clinical practice is a combination of advice, passive manual treatment techniques and neck exercises. The implementation of exercise for the treatment of chronic neck pain is indeed recommended in several clinical guidelines. Nevertheless, exercise programs show positive though limited effects, which can be explained by its biomechanical and physiological effects on muscles and joints, but a current lack of taking into account important biopsychosocial and neurophysiological factors. For instance, specific local exercises can lead to acute pain flare-ups, hampering patient satisfaction and the adherence to exercise programs. While it is shown that general aerobic exercise leads to decreased generalized pain sensitivity, also in the affected body parts, both immediately and on the longer term, although on the longer term the effects on local pain sensitivity are better for specific local exercises.

It can be hypothesized that a blended treatment program in which local specific neck exercises are combined with general aerobic exercise in counteractive amount will avoid pain flare-ups and maladaptive exercise perceptions, positively influencing treatment adherence and generating the most optimal clinical outcome due to the local and general effects.

Therefore the aim of this project is to investigate the effect of a blended treatment program (I) to a specific exercise program alone (C1) and to a general aerobic exercise program alone (C2) on pain intensity and cost effectiveness (primary outcome measures), and also on Global Perceived Effect, other pain-related outcomes, quality of life and functionality, lifestyle factors, and health-economic measures (secondary outcome measures) (O) in chronic non-specific neck pain patients (P).

ELIGIBILITY:
Inclusion Criteria:

* Neck pain > 3 months
* Mean pain intensity > 3/10 during the preceding month
* Native Dutch speaker
* Being able to walk normally

Exclusion Criteria:

* People with specific causes of neck pain (such as cervical disc herniation with nerve root impingement, severe osteoarthritis, fractures)
* Major depression or psychiatric illness
* Life threatening, metabolic, cardiovascular, neurologic, systemic diseases, diagnosed sleeping disorder
* Pregnancy or given birth in the preceding year
* History of head, neck or shoulder surgery
* Fibromyalgia and chronic fatigue syndrome
* Body mass index > 30 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | After treatment (12weeks)
  Pain intensity by the Brief Pain Inventory (BPI). The BPI includes four ratings of pain intensity (items 3-7), and seven other ratings on the impact of pain. Intensity is recorded on numerical scales from zero (no pain) to ten (pain as bad as you can imagine). Also, intensity is rated at the time of completing the questionnaires (pain now) as well as its worst, least, and average over the past day or week. The BPI also records the location of the pain on a diagram of a human figure. Patients are also asked to select words that best describe their pain and to indicate the extent and duration of pain relief obtained from analgesics.

SECONDARY OUTCOMES:
Pain sensitivity | Baseline and after 12 weeks treatment
  Pain sensitivity assessed by determine pressure pain thresholds (PPT) with an algometer at local and distal locations. Lower thresholds mean higher mechanical hypersensitivity.
Central sensitivity | Baseline and after 12 weeks treatment
  Central sensitivity by the Central Sensitization Inventory (CSI) questionnaire. The CSI is a two-part questionnaire that contains a 25-item survey that assesses the frequency of health-related symptoms associated with central sensitivity syndromes. Each question may be answered as follows:
  Never (0 points), Rarely (1 point), Sometimes (2 points), Often (3 points), or Always (4 points).
  The higher the total score, the more likely central sensitisation is present.
  Subclinical: 0 to 29 Mild: 30 to 39 Moderate: 40 to 49 Severe: 50 to 59 Extreme: 60 to 100
Pain intensity | baseline, after 6 weeks of treatment and 3 months after treatment
  Pain intensity by the Brief Pain Inventory (BPI). The BPI includes four ratings of pain intensity (items 3-7), and seven other ratings on the impact of pain. Intensity is recorded on numerical scales from zero (no pain) to ten (pain as bad as you can imagine). Also, intensity is rated at the time of completing the questionnaires (pain now) as well as its worst, least, and average over the past day or week. The BPI also records the location of the pain on a diagram of a human figure. Patients are also asked to select words that best describe their pain and to indicate the extent and duration of pain relief obtained from analgesics.
Neck pain-related disability | Baseline, after 6 weeks treatment, after 12 weeks treatment, after 3 months
  Neck pain-related disability assessed by the Neck Disability Index (NDI). The test has a maximum score of 50. 0 points means : no activity limitations , 50 points means complete activity limitation. A higher score indicates more patient-rated disability.
Health-related quality of life | Baseline, after 6 weeks treatment, after 12 weeks treatment, after 3 months
  Health-related quality of life assessed by the Short Form Health Survey- 36 items (SF-36).
  The questionnaire contains scales for physical and social function, mental health, energy, pain and general health perception. A higher score represents a better health.
Physical activity | Baseline and after 12 weeks of treatment
  Physical activity monitored by activity trackers.
Insomnia | Baseline and after 12 weeks treatment
  Self-reported sleep by the Insomnia Severity Index (ISI). The questionnaire assesses the severity of both nighttime and daytime components of insomnia. Scores are ranging from 0 to 28. The higher the score the worse the insomnia.
Sleep quality | Baseline and after 12 weeks treatment
  Sleep quality by the Pittsburgh Sleep Quality Index (PSQI). The PSQI-scores vary from 0 to 21. A score higher than 5 indicates bad sleep quality.
Stress | Baseline and after 12 weeks treatment
  Self-reported by the Depression Anxiety and Stress Scale (DASS). Participants indicate on a 4-point scale the extent to which each of 42 statements applied over the past week. Higher scores on each subscale indicate increasing severity of depression, anxiety, or stress.
Productivity losses | Baseline, after 6 weeks treatment, after 12 weeks treatment, after 3 months
  Productivity losses by iMTA Productivity Cost Questionnaire. The iMTA Productivity Cost Questionnaire (iPCQ) includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presenteeism and productivity losses related to 3) unpaid work.
Medical consumption | Baseline, after 6 weeks treatment, after 12 weeks treatment, after 3 months
  iMTA Medical Consumption Questionnaire (iMCQ), a generic instrument for measuring medical costs. The iMCQ includes questions related to frequently occurring contacts with health care providers.
Treatment adherence | Baseline, after 6 weeks treatment, after 12 weeks treatment, after 3 months
  The patient's ability to fully and accurately observe and perform the advice and instructions, will be evaluated by a online diary.
Global Perceived effect | Baseline, after 6 weeks treatment, after 12 weeks treatment, after 3 months
  The Global Perceived Effect (GPE) scale is a self-report tool for the patient to rate on a numeric scale, how much their pain condition has improved (+5) or worsened (-5) since a predefined time point.
Cost effectiveness | Baseline, after 6 weeks treatment, after 12 weeks treatment, after 3 months
  Euro Quality of life 5D questionnaire (score = 0-100, higher scores = better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Mira Meeus, Prof.Dr., Principal Investigator — University Ghent
Locations (1):
- Department of rehabilitation sciences (Ghent University), Ghent, Gente, Belgium